CLINICAL TRIAL: NCT03275090
Title: The Effects of Two Different Intravenous Lipid Emulsions on the Outcomes of Preterm Infants With Sepsis: a Randomized Pilot Controlled Trial
Brief Title: The Effects of Two Different Intravenous Lipid Emulsions on the Outcomes of Preterm Infants With Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Yahya Wahba, Principal Investigator, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MansouraUCH
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Sepsis Newborn
Keywords: lipid emulsions; preterm; sepsis
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth; Sepsis | interventions — SMOFlipid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralipid injectable product (MOFS) (Active Comparator): 20 preterm infants receive parenteral nutrition containing 20% MOFS lipid emulsion (Smoflipid ®)
  Interventions: Drug: Smoflipid ®
- Pure Soybean oil lipid emulsion (No Intervention): 20 preterm infants with sepsis receive the usual parenteral nutrition containing soybean oil based lipid emulsion (20% Intralipid ®) at daily increasing doses guided by serum triglycerides.

INTERVENTIONS:
Drug: Smoflipid ®
  Other Names: MOFS lipid emulsion
  Arms: Intralipid injectable product (MOFS)

SUMMARY:
Introduction and objectives: Lipid emulsions play an important role in parenteral nutrition in preterm infants. We aim to evaluate the effect of two different intravenous lipid emulsions on the outcomes of neonatal sepsis in preterm infants.

Methods: A randomized controlled trial is conducted in the Neonatal Care Unit of Mansoura University Children's Hospital, Egypt. Forty preterm infants with clinically suspected sepsis are enrolled and assigned randomly into one of two groups, one receive MOFS lipid emulsion (MOFS group) and the other receive pure soyabean oil-based emulsion (S group). Clinical and epidemiological data are collected. Assessment is done on 1st day and 7th day post randomization including growth parameters, complete blood count, C-reactive protein, random blood glucose, serum creatinine, serum triglyceride, soluble intercellular adhesion molecule 1 (sICAM-1) and leukocyte integrin β2. Between-groups and within-group differences will be analyzed statistically.

DETAILED DESCRIPTION:
1. Introduction Neonatal sepsis is a clinical syndrome of bacteremia with systemic symptoms and signs of infection in the first 28 days of life. In recent national studies, the incidence of suspected neonatal sepsis among admitted neonates varied from 32.9% to 45.9% with a higher incidence in preterm.

   Several soluble adhesion molecules are released in neonatal sepsis. Among these, soluble intercellular adhesion molecule 1 (sICAM-1) and leukocyte integrin β2 are early predictors of sepsis with high sensitivity and specificity.

   Septic preterm infants are more vulnerable to undernutrition and postnatal failure of growth requiring more nutritional support. The early use of adequate parenteral nutrition (PN) minimizes weight loss, improves growth and neurodevelopmental outcomes, and appears to reduce the risk of mortality. In preterm neonates, lipid emulsions (LE) play an important role in PN being an important source of energy, fat soluble vitamins and essential fatty acids. For the last few decades, pure soyabean oil based LE (S-LE) were used worldwide and consisted of long chain fatty acids with omega 3: omega 6 ratio of 1:5.5. Recently, LE preparations derived from multiple sources have been developed for clinical application. MOFS-LE mixture is one containing a mixture of 30% medium chain triglycerides (MCT), 25% olive oil, 15% fish oil, and 30% soyabean oil. They are supposed to have better immunomodulatory and anti-inflammatory properties with fewer side effects.

   There are several studies concerning the comparison between of S-LE and MOFS-LE as regards the efficacy and safety on neonates but without a consensus on the ideal LE .To our knowledge, this is the first randomized controlled trial (RCT) of two different intravenous LE conducted in septic preterm infants to unravel the short term effects of S-LE versus MOFS-LE on the outcomes of neonatal sepsis as well as on the serum levels of sICAM-1 and leukocyte integrin β2.
2. Materials and methods

2.1 Study design and participants Our study is a randomized controlled pilot trial that is conducted in the Neonatal Care Unit (NCU) of Mansoura University Children's Hospital, Egypt including 40 preterm infants. The study was accepted by International research board of Medical Faculty of Mansoura University.

Sepsis is defined clinically as the presence of three or more of the following groups of clinical signs: tachypnea (> 60 breath/min), retractions, nasal flaring, apnea, cyanosis; bradycardia (<100 beat/min), tachycardia (> 180 beat/min); seizures, hypotonia; poor skin color, capillary refill time > two seconds; lethargy, irritability.

2.2 Randomization Informed consents are obtained from the parents. Then, patients are assigned blindly into one of two groups using cards provided in opaque sealed consecutively numbered envelopes. MOFS group (n=20 cases) receive PN containing MOFS-LE which is a 30:30:25:15 mixture of soybean oil, MCT, olive oil, and fish oil (SMOFlipid ®, Fresenius kabi, Uppsala, Sweden) for seven consecutive days. S group (n=20 cases) receive PN containing S-LE (20% Intralipid ®, Fresenius kabi, Uppsala, Sweden) for seven consecutive days.

PN preparation is carried out by a special nurse under complete aseptic technique in a separate room and provided as (all in one) admixture. The all in one admixture is prepared daily following usual unit policy except for the type of intravenous LE and administrated through central venous catheters at a constant (pump controlled) rate for 24 hours per day. PN administration to preterm infants will be given according to the standard protocol of the unit. The starting dose of intravenous lipid is 0.5 g/kg/day on the first day of PN, increase gradually by 1gm/kg/day to a maximum dose of 3.5 gm/kg/day as recommended by the European Society for Clinical Nutrition and Metabolism (ESPEN)/European Society of Paediatric Gastroenterology, Hepatology, and Nutrition. As a rule, when serum triglyceride levels exceed 250 mg/dl, the lipid dosage will be reduced by 25% of the given dose. Amino acids, carbohydrates, trace elements, vitamins and electrolytes are given for both groups according to the unit's standard protocol.

Empirical antibiotics are started for the cases at the onset of clinically suspected sepsis according to our NCU policy. Cases of EOS receive ampicillin and gentamycin while cases of LOS receive with either cefotaxime or gentamycin.

2.3 Interventions Epidemiological and clinical data are collected including gestational age (assessed by early ultrasound scan, menstrual history and the new Ballard score), postnatal age, sex, birth weight, maternal age, type of delivery, risk factors for sepsis (maternal fever, urinary tract infection, prolonged rupture of membranes, central line insertion or surgical operation), duration of antibiotic treatment, mechanical ventilation, duration of hospital stay and mortality rate. Clinical examination is done on 1st day of suspicion of sepsis and seven days later including growth parameters (body weight, length and head circumference), vital signs, cardiovascular examination (skin perfusion and pulsations), chest examination (signs of respiratory distress and abnormal adventitious sounds), gastrointestinal system (abdominal distention, signs of feeding intolerance and organomegaly) as well as central nervous system examination (activity, neonatal reflexes, abnormal tone and seizures).

Laboratory investigations is done on 1st day of suspicion of sepsis and seven days post-randomization. Five ml of venous blood was withdrawn, 1 ml of them into Ethylene diamine tetra acetic acid (EDTA) tube for complete blood count (CBC), 1 ml blood into BACTEC vial for blood culture and 3 ml blood into a plain tube which was centrifuged and the resulting serum will be used for assay of C-reactive protein (CRP), random blood glucose, serum creatinine and serum triglyceride, sICAM-1 and leukocyte integrin ß2. Urine culture and cerebrospinal fluid examination will be done for LOS. Serum levels of sICAM-1 and leukocyte integrin ß2 are quantitatively measured by enzyme-linked immunosorbent assay (ELISA) technique.

2.4 Statistical analysis Statistical Package for the Social Sciences (SPSS) version 22 (IBM Corporation,Newyork, USA) was used to analyze data. Frequency (number and percent) will be used to express categorical variables. Chi square test is used for comparison of categorical variables between two groups. Fisher exact test is needed when more than 25% of the cells have expected count less than 5. Non-parametric data are presented as median and range, while parametric data are presented as mean ± standard deviation (SD). Between-groups comparisons are done using Student's t test (for parametric data) and Mann-Whitney test (for non-parametric data). Within-group comparisons of changes from 1st day to 7th day are carried out by means of Wilcoxon test for non-parametric data and paired t-test for parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 28 to less than 37 weeks who showed clinical symptoms and signs suggestive of early-onset sepsis (EOS, within 72 hours of birth) or late-onset sepsis (LOS, after 72 hours of birth) and received PN.

Exclusion Criteria: Neonates with

* Major congenital malformations
* Congenital heart diseases
* Inborn errors of metabolism
* Congenital infections
* Hypoxic-ischemic encephalopathy

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
levels of soluble intercellular adhesion molecule 1 (sICAM-1) | "first day of randomization and 7th days"
  changes in levels of sICAM-1 in septic preterm infants after receiving one of the two different lipid emulsions for seven days.
leukocyte integrin ß2 Level | "first day of randomization and 7th days"
  changes in leukocyte integrin ß2 level in septic preterm infants after receiving one of the two different lipid emulsions for seven days.

SECONDARY OUTCOMES:
duration of hospital stay | "through study completion, an average of 12 months"
  Effect of two different lipid emulsions on hospital stay duration in septic preterm infants
Duration of antibiotic treatment | "through study completion, an average of 12 months"
  Effect of two different lipid emulsions on duration of antibiotics treatment in septic preterm infants
Duration of mechanical ventilation | "through study completion, an average of 12 months"
  Effect of two different lipid emulsions on duration of mechanical ventilation in septic preterm infants
Mortality rate | "through study completion, an average of 12 months"
  Effect of two different lipid emulsions on mortality rate in septic preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Yahya M Wahba, MD, Principal Investigator — Mansoura University Children Hospital
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paolucci M, Landini MP, Sambri V. How can the microbiologist help in diagnosing neonatal sepsis? Int J Pediatr. 2012;2012:120139. doi: 10.1155/2012/120139. Epub 2012 Jan 26. PMID 22319539
- [Result] Mohsen L, Ramy N, Saied D, Akmal D, Salama N, Abdel Haleim MM, Aly H. Emerging antimicrobial resistance in early and late-onset neonatal sepsis. Antimicrob Resist Infect Control. 2017 Jun 13;6:63. doi: 10.1186/s13756-017-0225-9. eCollection 2017. PMID 28630687
- [Result] Shehab El-Din EM, El-Sokkary MM, Bassiouny MR, Hassan R. Epidemiology of Neonatal Sepsis and Implicated Pathogens: A Study from Egypt. Biomed Res Int. 2015;2015:509484. doi: 10.1155/2015/509484. Epub 2015 Jun 4. PMID 26146621
- [Result] Edgar JD, Gabriel V, Gallimore JR, McMillan SA, Grant J. A prospective study of the sensitivity, specificity and diagnostic performance of soluble intercellular adhesion molecule 1, highly sensitive C-reactive protein, soluble E-selectin and serum amyloid A in the diagnosis of neonatal infection. BMC Pediatr. 2010 Apr 16;10:22. doi: 10.1186/1471-2431-10-22. PMID 20398379
- [Result] Mishra UK, Jacobs SE, Doyle LW, Garland SM. Newer approaches to the diagnosis of early onset neonatal sepsis. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F208-12. doi: 10.1136/adc.2004.064188. PMID 16632649
- [Result] Turunen R, Andersson S, Nupponen I, Kautiainen H, Siitonen S, Repo H. Increased CD11b-density on circulating phagocytes as an early sign of late-onset sepsis in extremely low-birth-weight infants. Pediatr Res. 2005 Feb;57(2):270-5. doi: 10.1203/01.PDR.0000148717.59861.2C. Epub 2004 Dec 7. PMID 15585684
- [Result] Ramel SE, Brown LD, Georgieff MK. The Impact of Neonatal Illness on Nutritional Requirements-One Size Does Not Fit All. Curr Pediatr Rep. 2014 Dec;2(4):248-254. doi: 10.1007/s40124-014-0059-3. PMID 25722954
- [Result] Christmann V, Visser R, Engelkes M, de Grauw AM, van Goudoever JB, van Heijst AF. The enigma to achieve normal postnatal growth in preterm infants--using parenteral or enteral nutrition? Acta Paediatr. 2013 May;102(5):471-9. doi: 10.1111/apa.12188. Epub 2013 Feb 25. PMID 23398476
- [Result] Kapoor V, Glover R, Malviya MN. Alternative lipid emulsions versus pure soy oil based lipid emulsions for parenterally fed preterm infants. Cochrane Database Syst Rev. 2015 Dec 2;2015(12):CD009172. doi: 10.1002/14651858.CD009172.pub2. PMID 26630252
- [Result] de Meijer VE, Gura KM, Le HD, Meisel JA, Puder M. Fish oil-based lipid emulsions prevent and reverse parenteral nutrition-associated liver disease: the Boston experience. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):541-7. doi: 10.1177/0148607109332773. Epub 2009 Jul 1. PMID 19571170
- [Result] Koletzko B, Goulet O. Fish oil containing intravenous lipid emulsions in parenteral nutrition-associated cholestatic liver disease. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):321-6. doi: 10.1097/MCO.0b013e3283385407. PMID 20393276
- [Result] Resch B, Gusenleitner W, Muller WD. Procalcitonin and interleukin-6 in the diagnosis of early-onset sepsis of the neonate. Acta Paediatr. 2003;92(2):243-5. doi: 10.1111/j.1651-2227.2003.tb00534.x. PMID 12710654
- [Result] Koletzko B, Goulet O, Hunt J, Krohn K, Shamir R; Parenteral Nutrition Guidelines Working Group; European Society for Clinical Nutrition and Metabolism; European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN); European Society of Paediatric Research (ESPR). 1. Guidelines on Paediatric Parenteral Nutrition of the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) and the European Society for Clinical Nutrition and Metabolism (ESPEN), Supported by the European Society of Paediatric Research (ESPR). J Pediatr Gastroenterol Nutr. 2005 Nov;41 Suppl 2:S1-87. doi: 10.1097/01.mpg.0000181841.07090.f4. No abstract available. PMID 16254497
- [Result] Al-Taiar A, Hammoud MS, Cuiqing L, Lee JK, Lui KM, Nakwan N, Isaacs D. Neonatal infections in China, Malaysia, Hong Kong and Thailand. Arch Dis Child Fetal Neonatal Ed. 2013 May;98(3):F249-55. doi: 10.1136/archdischild-2012-301767. Epub 2012 Aug 31. PMID 22942104